CLINICAL TRIAL: NCT00004094
Title: A Phase II Study of Induction Chemotherapy Followed by Concomitant Paclitaxel (1 Hour Infusion), Fluorouracil, Hydroxyurea and Hyperfractionated Radiotherapy for Advanced Oral, Pharynx and Larynx Cancer
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Previously Untreated Advanced Cancer of the Mouth, Pharynx, or Larynx
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: University of Chicago
Purpose: Treatment
Other Study IDs: NU C98N1; NU-C98N1; UCCRC-9502; NCI-G99-1587
Record Dates: First submitted 1999-12-10; First posted 2003-05-08 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-12

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Fluorouracil; Hydroxyurea; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: fluorouracil
Drug: hydroxyurea
Drug: paclitaxel
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have previously untreated advanced cancer of the mouth, pharynx, or larynx.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the activity of induction chemotherapy with carboplatin and paclitaxel followed by concurrent fluorouracil, hydroxyurea, paclitaxel, and hyperfractionated radiotherapy in terms of response rate, pattern of failure, time to progression, and overall survival in patients with previously untreated advanced oral, pharyngeal, or laryngeal cancer.
* Assess this treatment regimen in terms of the pattern and degree of clinical acute, cumulative, and chronic toxic effects in this patient population.
* Assess the rate of organ preservation in resectable patients treated with this regimen.
* Evaluate the quality of life, organ function, and incidence of second primary tumors in patients treated with this regimen.
* Assess the rate of complications with subcutaneously implanted IV infusion catheters in patients treated with this regimen.

OUTLINE: Patients receive induction chemotherapy comprising paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes weekly for 3 weeks. Treatment repeats every 4 weeks for 2 courses.

At 1-2 weeks after completion of induction chemotherapy, patients receive oral hydroxyurea every 12 hours on days 1-6, fluorouracil IV continuously on days 1-5, radiotherapy twice daily on days 1-5, and paclitaxel IV over 1 hour on day 2. Treatment repeats every 2 weeks for 5 courses.

Patients with residual nodal disease or initially staged nodal disease in the absence of macroscopic residual disease undergo neck dissection after completion of chemoradiotherapy. Patients with residual disease at the primary site undergo complete excision of disease. Patients with disease progression or disease recurrence are considered for conventional surgical management.

Quality of life is assessed every 3 months for 6 months, every 6 months for 1.5 years, and then annually thereafter.

Patients are followed monthly for 1 year, every 2 months for 1 year, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell or poorly differentiated carcinomas, or lymphoepithelioma of the head and neck

  * Stage III carcinoma of the base of the tongue or hypopharynx
  * Stage IV carcinoma of the oral cavity, pharynx (including nasopharynx, oropharynx, and hypopharynx), or larynx
* No distant metastasis
* Measurable disease desirable

  * Clinically disease free after prior surgery allowed

PATIENT CHARACTERISTICS:

Age:

* 15 to 80

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No clinically significant cardiomyopathy or congestive heart failure

Pulmonary:

* No clinically significant pulmonary dysfunction

Other:

* No severe baseline neurologic deficits
* No uncontrolled active infection other than that not curable without treatment of cancer
* No sensitivity to Cremophor EL
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics
* Incisional or excisional biopsy and organ sparing procedures (e.g., debulking of airway compromising tumors or neck dissection) in patients with an existing primary tumor allowed
* No more than 3 months since prior nonbiopsy procedure

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (4):
- United States (4):
  - Monroe Medical Associates, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois